CLINICAL TRIAL: NCT01957007
Title: A Phase 1b Study of Vantictumab (OMP-18R5) in Combination With Docetaxel in Patients With Previously Treated Non-Small Cell Lung Cancer
Brief Title: A Study of Vantictumab (OMP-18R5) in Combination With Docetaxel in Patients With Previously Treated NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18R5-004
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors
Keywords: Phase 1; dose escalation; histologically confirmed; malignancy metastatic
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Experimental): Drug: Docetaxel - administered intravenously
  Interventions: Drug: Docetaxel; Drug: vantictumab
- vantictumab (Experimental): Drug: vantictumab - administered intravenously
  Interventions: Drug: Docetaxel; Drug: vantictumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be administered IV.
Drug: vantictumab — Vantictumab will be administered intravenously
  Other Names: (OMP-18R5)

SUMMARY:
This is an open-label Phase 1b dose-escalation study to assess the safety, tolerability, and PK of vantictumab when combined with docetaxel.

DETAILED DESCRIPTION:
Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined, up to 10 patients may be enrolled in the cohort-expansion phase to better characterize the safety, tolerability and PK of vantictumab combined with docetaxel. Up to approximately 34 patients may be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Histologically documented recurrent or advanced (Stage IV) NSCLC
* Eastern CooperativeOncology Group (ECOG) performance status of 0 or 1
* All acute treatmentrelated toxicity from prior therapy must have resolved to Grade ≤ 1 prior to study entry
* Adequate hematologic and end-organ function
* Evaluable or measurable disease per RECIST v1.1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

* Prior treatment with docetaxel for recurrent or advanced NSCLC
* More than two regimens of systemic cytotoxic chemotherapy for recurrent or advanced NSCLC
* Treatment with any anti-cancer therapy within 3 weeks prior to initiation of study treatment
* Known hypersensitivity to any component of study treatments
* Grade ≥ 2 sensory neuropathy
* Uncontrolled seizure disorder or active neurologic disease
* Untreated brain metastases
* Leptomeningeal disease as a manifestation of cancer
* Active infection requiring antibiotics
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known history of clinically significant liver disease, including active viral hepatitis and cirrhosis
* Significant intercurrent illness including, but not limited to, unstable angina pectoris, and cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnancy, lactation, or breastfeeding
* Known HIV infection
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Concurrent use of therapeutic warfarin
* New York Heart Association Classification III or IV (see Appendix E)
* Known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of study treatment or anticipation of need for major surgical procedure during the course of the study
* Osteoporosis based on a T-score of <-2.5 at the left or right total hip, left or right femoral neck or lumbar spine (L1-L4) as determined by DEXA scan
* Bone metastases and one of the following:

  * Prior history of a pathologic fracture
  * Lytic lesion requiring an impending orthopedic intervention
  * Lack of treatment with a bisphosphonate or denosumab
* Treatment with a thiazolidinedione PPAR gamma inhibitor; e.g. Actos® (pioglitazone), and Avandia® (rosiglitzone)
* Active treatment with an oral or IV glucocortocoid for ≥4 weeks at a daily dose equivalent to or greater than 7.5 mg of oral prednisone
* Fasting β-CTX of >1000 pg/mL
* Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of vantictumab in combination with docetaxel in patients with recurrent or advanced NSCLC. The maximum tolerated dose (MTD) will be determined in patients treated with vantictumab in combination with weekly paclitaxel. | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-28)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of vantictumab when administered in combination with docetaxel to patients with recurrent or advanced NSCLC | Plasma sample for Pharmacokinetics (PK) analysis to be obtained prior to the vantictumab infusion and before docetaxel infusion from Day 0 to treatment termination
  Apparent half life, AUC, clearance, volume of distribution

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - Roswell Park Cancer Center, Elm & Carlton Streets, Buffalo, New York
  - Case Western Reserve University, Cleveland, Ohio